CLINICAL TRIAL: NCT00865163
Title: LASER: Real Life Antithrombotic Stent Evaluation Registry
Acronym: LASER
Status: Completed | Type: Observational
Sponsor: Stiftung Institut fuer Herzinfarktforschung (Other)
Responsible Party: Sponsor
Other Study IDs: LASER Registry
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Percutaneous Coronary Intervention
Keywords: Percutaneous Coronary Intervention; anticoagulation; PCI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
LASER is designed to gather data about ischemic an bleeding complications for a period of 12 months after a PCI with the aim to optimize the therapy of these patients.

DETAILED DESCRIPTION:
The LASER Registry will collect data from unselected patients on how the problem of stents on the background of full anticoagulation is approached by the investigators. On the collected data the LASER registry will

* document the frequently used treatment modalities how patients requiring stents on the background of full anticoagulation with Vitamin K Antagonists are currently managed
* will document the associated cardiac event rates with each currently used treatment strategy
* will document the associated bleeding rates with each currently used treatment strategy

With these data available, the LASER Registry will allow

* to define an optimised treatment regimen for the treatment of patients on full anticoagulation with Vitamin K Antagonists receiving one or more coronary stents
* to allow the appropriate sample size calculation for the design of a subsequent randomised comparison of continuous triple anticoagulation versus this optimised treatment regimen in such patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with significant symptomatic coronary artery disease (stable angina class II or more (CCS) , unstable angina, NSTEMI, or STEMI) and who for this reason do undergo percutaneous coronary revascularization with one or more drug eluting stent(s) (DES) or bare metal stent(s)
* Patients requiring Vitamin K Antagonists based full anticoagulation therapy (target INR 2-4,5) for any clinical indication
* Age: >18 years; no upper age limit
* Informed consent has been obtained that the patient agrees to be fol-lowed up for up to one year

Exclusion Criteria:

* Patients who have been treated with a combined anticoagulant & antiplatelet therapy within the previous two months
* Overt or constant occult bleeding that cannot adequately be treated (proton pump inhibitors, H2-blockers e.g.)
* Any contraindication to the use of thienopyridines
* Any contraindication to the use of aspirin
* Severe liver or kidney disease
* Any reason that creates sufficient doubts that follow-up can be obtained with reasonable efforts
* Any other reason that in the eye of the investigator makes the patient unsuitable for the participation in the registry
* For female patients only: pregnant or not on oral contraceptives or child bearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with significant symptomatic coronary artery disease who for this reason undergo PCI with implantation of one or more drug eluting stent(s) (DES) or bare metal stent(s) and requiring Vitamin K Antagonist based full anticoagulation therapy (target INR 2-4,5) for any clinical indication.
  The LASER Registry will collect the data of 1000 patients with the need for oral anticoagulation and 1000 matched control patients without the need for oral anticoagulation.
Sampling Method: Non-Probability Sample
Enrollment: 915 (Actual)
Dates: Start 2008-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dietrich C. Gulba, MD, Principal Investigator — Krankenhaus Düren
Locations (2):
- Germany (2):
  - Krankenhaus Düren, Düren
  - Institut für Herzinfarkforschung Ludwigshafen, Ludwigshafen

IPD SHARING:
Plan to Share IPD: No